CLINICAL TRIAL: NCT01813591
Title: A Randomized, Open-Label, Parallel Two-Arm Study Evaluating the Efficacy of H.P. Acthar Injection Gel in the Treatment of Adults With Intractable Chronic Migraine
Brief Title: A Two-Arm Study Evaluation H.P. Acthar Injection Gel in Treatment of Chronic Migraines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dent Neuroscience Research Center (Other)
Responsible Party: Principal Investigator, Laszlo L. Mechtler, M.D., Chief Medical Officer, Dent Neuroscience Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTHAR
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Chronic Migraine
Keywords: Chronic Migraine; Headache; Refractory Chronic Migraine
MeSH Terms: conditions — Headache | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- H.P. Acthar Gel 80IU (Experimental): H.P. Acthar Gel of 80IU (1.0 ml)
  Interventions: Drug: H.P. Acthar Gel
- H.P. Acthar Gel 40IU (Experimental): H.P. Acthar Gel of 40IU (0.5 mL)
  Interventions: Drug: H.P. Acthar Gel

INTERVENTIONS:
Drug: H.P. Acthar Gel — Acthar (40IU or 80IU) given subcutaneously for 5 days in the 1st week, followed by every other day (3 times per week for the next 3 weeks)
  Other Names: Acthar; Repository Corticotropin Injection; ACTH Gel

SUMMARY:
This small study is to investigate the efficacy of Acthar in the treatment of chronic migraine in patients who have failed multiple treatments, including Botox (which is defined as having <30% reduction from baseline in the number of headache days per month). Despite the widespread use of anti-seizure medications, there remain a significant number of patient whose migraines are refractory to these agents. The pathophysiology of migraine is such that the neural substances calcitonin G related protein (CGRP), substance P, and neurokinin A are released at the trigeminal nerve endings innervating the large cranial and dura mater blood vessels and this neurotrasmission generates migraine associated pain. Because of this, treatment for migraine can be directed towards down regulating those receptor sites accordingly. Acthar may provide pain relief through this mechanist, as ACTH has been shown to inhibit the release of CGRP and may also provide relief through a negative feedback loop as exogenous ACTH inhibits CRH release and mast cell degranulation.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female, 18 to 60 years of age.
* Has a history of chronic migraine as classified by the International Headache Classification, ICHD-2R (i.e. must demonstrate an average of >=15 headache days per month, of which >=8 must be migraine days or >=8 days of migraine-specific acute medication-ergotamine or triptans for at least 3 months prior to study.
* Must demonstrate at least >=8 migraine days or >=8 days of migraine specific acute medications- ergotamine or triptans during 30 day baseline screening.
* Is able to differentiate migraine from any other headache they may experience (e.g., tension-type headache).
* Will have a previous history of failing at least one prophylactic treatment, which can include anti-seizure medications and/or TCA's prescribed for the treatment of chronic migraine.
* Must be considered a non-responder to previous treatment with Botox. Botox failure will be defined by previous documentation (at the discretion of the PI) or as having less than 30% reduction of headache days per month on Botox.
* Will have not had botulinum toxin with in 4 months before study enrollment.
* If female of childbearing potential, will have a negative urine pregnancy test at Visits 1 and 7, and uses, or agrees to use, for the duration of the study, a medically acceptable form of contraception as determined by the investigator.

  1. Complete abstinence from intercourse from 2 weeks prior to administration of study drug throughout the study, and for a time interval after completion or premature discontinuation from the study to account for elimination of the study drug (a minimum of 7 days); or,
  2. Surgically sterile (hysterectomy or tubal ligation or otherwise incapable of pregnancy); or,
  3. Sterilization of male partner; or,
  4. Intrauterine device with published data showing lowest expected failure rate is less than 1% per year; or,
  5. Double barrier method (i.e., 2 physical barriers OR 1 physical barrier plus spermicide) for a least 1 month prior to Visit 1 and throughout study; or,
  6. Hormonal contraceptives for at least 3 months prior to Visit 1 and throughout study. Protocol Number/v.1/06 Jun 2012 7
* Must be in generally good health as confirmed by medical history, baseline physical exam, baseline neurological exam and vital signs.

Exclusion Criteria:

* Is unable to understand the study requirements, the informed consent, or complete headache records as required per protocol.
* Is pregnant, actively trying to become pregnant, or breast-feeding.
* Has a significant systemic disease that is equally painful or more painful than migraine.
* Has a progressive neurological disorder such as MS.
* Has a history of chronic disease of the immune system other than MS or a known immunodeficiency syndrome such as HIV.
* Has sensitivity to proteins of porcine origin.
* Has a known or 'new' diagnosis of diabetes mellitus (if screening blood glucose is suspicious for diabetes [> or equal to 126 mg/dL or > or equal to 7 mmol/L if fasting;> or equal to 200 mg/dL or 11.1 mmol/L if random testing] a patient should be further evaluated for diabetes mellitus), or a known or 'new' diagnosis of hypothyroidism not adequately controlled with medication.
* Has previously taken Acthar for any reason.
* Has any contraindications listed on the Acthar PI.
* Has a history of cluster headache, chronic tension type headache, or headache due to medication over use according to IHS guidelines, in the 3 months prior to study enrollment or during the baseline phase.
* Has received any other investigative drug 30 days prior to enrollment in this study.
* Who in the opinion of the Principal Investigator has a condition for which they should not be enrolled in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Average total number of headache days (both 40IU and 80IU groups) | After 30 days of treatment
  Comparison of the average total number of headache days after 30 days of Acthar treatment (both 40IU and 80IU groups)with the average number of headache days at baseline screening period

SECONDARY OUTCOMES:
Total number of headache days (both 40IU and 80IU groups) | After 30 days of treatment
  Comparison of the total number of headache days after 30 days of Acthar treatment (both 40IU and 80IU groups) with the number of headache days at baseline screening period

OTHER OUTCOMES:
Number of headache and migraine days for a 40IU group | After 30 days of treatment
  A hierarchical analysis of the number of headache and (separately) migraine days subjects on 40IU experience on average during the 30 day treatment period compared to the number they experienced on average during the baseline screening period. If statistical significance (p<.05) is reached, then the 80IU subjects will be analyzed similarly

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo L Mechtler, M.D., Principal Investigator — Dent Neurologic Institute; John F Rothrock, M.D., Principal Investigator — Renown Institute for Neurosciences; Roger K Cady, M.D., Principal Investigator — Clinvest; Frederick G Freitag, M.D., Principal Investigator — Baylor Health Care System
Locations (4):
- United States (4):
  - Clinvest/A Division of Banyan Group, Inc., Springfield, Missouri
  - Renown Institute of Neurosciences, Reno, Nevada
  - Dent Neurologic Institute, Amherst, New York
  - Baylor University Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided